BERKELEY DAVIS IRVINE LOS ANGELES MERCED RIVERSIDE SAN DIEGO



SAN FRANCISCO SANTA BARBARA SANTA CRUZ

9500 GILMAN DRIVE, MC 0725 LA JOLLA, CALIFORNIA 92093-0725

HERBERT WERTHEIM SCHOOL OF PUBLIC HEALTH and HUMAN LONGEVITY SCIENCE

MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making

Principal Investigator: Andrea LaCroix, PhD
UC San Diego
Herbert Wertheim School of Public Health and Human Longevity Science
Email: alacroix@ucsd.edu

NCT: 05299983 Study Protocol: 3/31/2023

# MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making

## **Study Protocol**

#### **Study Participants**

Participants will meet the following eligibility criteria:

- Age 40 60 years
- Reside in the U.S.
- Have questions about their own perimenopause/menopause or at least one symptom
- Have interest in looking at a website about menopause for themselves
- Willingness to spend at least 20 minutes on a website and answer a 15-minute questionnaire
- Able to read and write in English

### **Recruitment & Informed Consent**

The study has approval by the Institutional Review Board at the University of California, San Diego Human Research Protections Program Office, (140604) and registered at the Clinical Trial Registry www.clinicaltrials (NCT05299983).

Participants will be recruited nationally using IRB approved advertisements on Facebook & Instagram. Once a participant clicks on a Facebook or Instagram ad, an online form in Qualtrics will open. Participants will read the information sheet (consent) and provide online consent. Participants will need to provide an email address. Once a participant provides consent, they will immediately receive an email with the study link. After opening the survey, the participants will complete a demographics survey and then will be randomized to one of two study groups (See **Study Design** below).

#### **Study Design**

Participants will be randomized to one of two study groups and be asked to leave the survey open, spend at least 20 minutes on the website(s), and then return to complete the survey:

- MyMenoPlan (Intervention group)
  - o Participants will review the MyMenoPlan.org website
- Control
  - Participants will be able to view any website of their choice including three high quality websites linked in the survey that were run by scientific, noncommercial, or governmental orgs.
    - https://www.menopause.org/for-women
    - https://www.womenshealth.gov/menopause
    - https://www.nia.nih.gov/health/topics/menopause

Compensation – Participants will receive \$30 if they passed all fraud detection (see below) and completed all the study tasks.

#### Fraud detection and noncompliance

One difficulty with studies that are conducted entirely only online is that there is an opportunity for bots, bad actors, and others who are not eligible to attempt to complete the study for the incentive money. We will employ the following fraud detection and noncompliance quality checks:

- Include the requirements for payment listed on information sheet, so that we can eliminate and not pay people who did not meet the inclusion criteria.
- The survey software will use reCAPTCHA to detect and eliminate bots.
- Eliminate participants who:
  - o spend less than 30 minutes combined on the site and questionnaire,
  - put in straight-lined responses to significant portions of the survey (giving the same answer across a large sequence of questions, despite reverse coded items)
  - fail attention checks (not giving the requested answer to an item on the survey like "Select answer B for this question").
- Not allow more than one survey completion from the same IP or email address.
  - We will manually check the consistency of names, addresses, phones, and email addresses at Spokeo.com, an online people look-up service.

#### Measures

Primary Outcome Measures:

- Perceived Quality of Information
  - This 7-item, 5-point Likert scale (1- Strongly disagree to 5 Strongly agree) is adapted from the Post-Study System Usability Questionnaire (PSSUQ) in Lewis (1995).
- Readability
  - This 2-item, 5-point Likert (1- Strongly disagree to 5 Strongly agree)scale was derived from the Standardized User Experience Percentile Rank Questionnaire (SUPR-Q) in Sauro (1995).
- Self-Efficacy for Managing Menopause Symptoms
  - This is a newly developed Likert scale (1- Strongly disagree to 5 Strongly agree) for assessing participants' beliefs in their own abilities in managing menopausal symptoms.
- Credibility
  - This 2-item, 5-point Likert (1- Strongly disagree to 5 Strongly agree) scale was derived from the Standardized User Experience Percentile Rank Questionnaire (SUPR-Q) in Sauro (1995).